CLINICAL TRIAL: NCT02950558
Title: Pilot Study: Extended Regional Anesthesia to Prevent Chronic Pain After Ankle Fracture Surgery
Brief Title: Anesthesia for Pain After Ankle Fracture Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Jun-ming Zhang, Professor of Anesthesia, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zhang2016
Record Dates: First submitted 2016-10-04; First posted 2016-11-01 (Estimated); Results first posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Chronic Pain; Ankle Fracture Surgery; Regional Anesthesia
MeSH Terms: conditions — Chronic Pain | interventions — Ropivacaine; Nerve Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ropivacaine (Active Comparator): Single injection of ropivacaine immediately prior to surgery
  Interventions: Drug: Ropivacaine
- Ropivacaine plus Nerve Block (Experimental): Single injection of ropivacaine immediately prior to surgery plus 5 day ambulatory popliteal nerve block.
  Interventions: Drug: Ropivacaine; Procedure: Nerve block

INTERVENTIONS:
Drug: Ropivacaine — Single injection of ropivacaine immediately prior to surgery.
  Other Names: Naropin
Procedure: Nerve block — insertion of catheter to deliver continuous 5 day popliteal sciatic nerve block using a disposable ambulatory pain pump.
  Other Names: no other name
  Arms: Ropivacaine plus Nerve Block

SUMMARY:
This pilot study will test the hypothesis that prolonged regional peripheral nerve block will reduce development of chronic pain in patients undergoing surgery for ankle fracture compared to standard of care. Subjects will be followed for one year.

DETAILED DESCRIPTION:
This pilot study will test the hypothesis that prolonged regional peripheral nerve block will reduce development of chronic pain in patients undergoing surgery for ankle fracture. Regional nerve block using local anesthetics delivered by ambulatory pump is used in some types of surgeries but is not routine for ankle fracture patients in our hospitals. Patients will be randomized to standard care (single shot peripheral nerve block prior to surgery) or experimental (the same single shot nerve block, followed by continuous popliteal nerve block with ropivacaine starting just after surgery). The primary outcome will be scores on a validated ankle/foot pain questionnaire that includes questions on function. Subjects will be followed for one year. Secondary outcome will be postoperative opioid use.

ELIGIBILITY:
Inclusion Criteria:

* Referred for surgery for open reduction and internal fixation for ankle fracture

Exclusion Criteria:

* Unable to give informed consent in English
* Unable to complete surveys in English
* Unable to understand instructions for using pump in English
* Unavailable for followup
* Polytrauma; undergoing other surgeries or having other orthopedic injuries related to the precipitating cause of the ankle fracture
* Infection
* Peripheral vascular disease
* Diabetes
* Currently undergoing chemotherapy
* Pregnancy
* Currently lactating
* Heart disease or heart rhythm disorder or taking anti-arrhythmic drugs
* Severe renal impairment (Class 3 or worse kidney disease)
* Liver disease (cirrhosis or liver failure)
* Prior allergic reaction to any type of local anesthetic
* Taking therapeutic doses of anti-coagulants or anti-platelet therapy (prophylactic doses started because of hospital admission are not an exclusion)
* Currently taking antidepressants or other psychiatric medications
* Single shot local nerve block prior to surgery was ineffective
* Selected for neuraxial anesthesia rather than general anesthesia for the open reduction surgery
* Already receiving chronic analgesic therapy for a separate chronic pain condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2020-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Ming Zhang, MD, MSc, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - UC Health West Chester Hosptial, West Chester, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients scheduled for open reduction and fixation of an ankle fracture were recruited from hospitals and outpatient surgery centers associated with the University of Cincinnati. Recruitment was delayed by a national ropivacaine shortage. Recruitment occurred between May 2018 and June 2019.
Groups:
- Standard Care: Single injection of ropivacaine immediately prior to surgery
  Ropivacaine: Single injection of ropivacaine immediately prior to surgery.
- Ropivacaine Pump: Single injection of ropivacaine immediately prior to surgery plus 5 day ambulatory popliteal nerve block.
  Ropivacaine: Single injection of ropivacaine immediately prior to surgery.
  Nerve block: insertion of catheter to deliver continuous 5 day popliteal sciatic nerve block using a disposable ambulatory pain pump.
Period: Overall Study
Arm/Group | Standard Care | Ropivacaine Pump
Started | 8 | 6
12 Month Pain Questionnaire | 6 | 6
Completed | 6 | 6
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Ropivacaine Pump | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.13 (10.09) | 43.17 (15.41) | 43.71 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 6 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 14
BMI (body mass index) [Mean (Standard Deviation); unit: kg/m^2] | 31.17 (5.538) | 31.53 (3.886) | 31.32 (4.728)

OUTCOME MEASURES:

1. Primary Outcome: Pain Score at 12 Months - Experimental Group vs. Control Group
Description: Patients will complete Self-Administered Foot and Ankle Questionnaire (SEFAS) at 12 months post surgery. 0 = worst possible pain and function, 48 = no pain or dysfunction. Higher scores indicate a better outcome.
Time Frame: at 12 months post surgery
Population: 2 subjects in standard care group were lost to follow-up and did not complete 12 month questionnaire but their questionnaires from earlier time points were included in the analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | Ropivacaine Pump
Number analyzed (Participants) | 6 | 6
units on a scale | 36.33 (9.543) | 44.00 (1.414)
Statistical Analysis 1: Comparison: Standard Care vs Ropivacaine Pump; Test type: Other; p = 0.1269, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Pain Score at 2 Weeks - Experimental Group vs. Control Group
Description: Patients will complete Self-Administered Foot and Ankle Questionnaire at 2 weeks post surgery. For this instrument, 0 = worst possible pain and function, 48 = no pain or dysfunction. Higher scores indicate a better outcome
Time Frame: at 2 weeks post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | Ropivacaine Pump
Number analyzed (Participants) | 8 | 6
units on a scale | 16.22 (6.637) | 13.67 (2.082)
Statistical Analysis 1: Comparison: Standard Care vs Ropivacaine Pump; Test type: Other; p = 0.8808, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Pain Score at 3 Months - Experimental Group vs. Control Group
Description: Patients will complete Self-Administered Foot and Ankle Questionnaire at 3 months post surgery. 0 = worst possible pain and function, 48 = no pain or dysfunction. Higher scores indicate a better outcome.
Time Frame: at 3 months post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | Ropivacaine Pump
Number analyzed (Participants) | 8 | 6
units on a scale | 26.25 (7.869) | 35.71 (5.489)
Statistical Analysis 1: Comparison: Standard Care vs Ropivacaine Pump; Test type: Other; p = 0.0382, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Pain Score at 6 Months - Experimental Group vs. Control Group
Description: Patients will complete Self-Administered Foot and Ankle Questionnaire at 6 months post surgery. 0 = worst possible pain and function, 48 = no pain or dysfunction. Higher scores indicate a better outcome.
Time Frame: at 6 months post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ropivacaine Ppump: Single injection of ropivacaine immediately prior to surgery plus 5 day ambulatory popliteal nerve block.
  Ropivacaine: Single injection of ropivacaine immediately prior to surgery.
  Nerve block: insertion of catheter to deliver continuous 5 day popliteal sciatic nerve block using a disposable ambulatory pain pump.
Arm/Group | Standard Care | Ropivacaine Ppump
Number analyzed (Participants) | 6 | 6
units on a scale | 34.00 (9.011) | 37.67 (3.724)
Statistical Analysis 1: Comparison: Standard Care vs Ropivacaine Ppump; Test type: Other; p = 0.4696, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Incidence of Chronic Ankle Pain Diagnoses - Experimental Group vs. Control Group
Description: Incidence of chronic ankle pain diagnoses one year after surgery obtained from the medical record was originally planned but proved difficult to obtain. Here we provide the number of patients with a 12 month Self-Administered Foot and Ankle Questionnaire score lower than 40 at the 12 month time point. For this instrument, 48 = no pain or disability; 0 = maximum pain and disability. Scores of 40 below were interpreted to indicate ongoing ankle pain of significance for pain and function, for example, at least 8 of the 12 questions being scored less than the optimal value of 4. Scores from 40 to 48 were interpreted as indicating normal or near normal function of the affected ankle.
Time Frame: at 1 year post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Ropivacaine Pump
Number analyzed (Participants) | 6 | 6
Participants
  SEFAS Score >=40 | 3 | 6
  SEFAS Score <40 | 3 | 0
Statistical Analysis 1: Comparison: Standard Care vs Ropivacaine Pump; Test type: Other; p = 0.1818, Fisher Exact

ADVERSE EVENTS:
Time Frame: Subjects were contacted daily by phone for the first five days after surgery (which corresponded to the duration of ambulatory ropivacaine pump use for subjects in the experimental group). Medical chart records were reviewed for adverse events for 3 months following the surgery.
Description: The protocol incorporated FDA adverse event definitions and Good Clinical Practices.
Arm/Group | Standard Care | Ropivacaine Pump
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 1/8 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=8) | Ropivacaine Pump (N=6)
wound dehiscence (Surgical and medical procedures) | 1 (1) | 0 (0)
metalic taste around lips (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lightheadedness, nausea,headache (General disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
A problem encountered was that only 1 of the 6 subjects in the pump group received the full 5 days of treatment. The others discontinued using the pump early, primarily due to problems with catheter dislodgement/leakage. As specified in the statistical analysis plan, these subjects were all analyzed with intent-to-treat protocol and are included in the pump group data presented. Also, by chance, the distribution of males and females between the group was quite uneven.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT02950558/Prot_001.pdf
  • Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT02950558/SAP_000.pdf